CLINICAL TRIAL: NCT06400654
Title: Retrospective and Prospective Observational Study on prognostIc and Predictive Factors in Patients With Extra-pulmonary, adVanced Neuroendocrine cArciNomas and Mixed Adeno-neuroendocrine Carcinomas (NIRVANA)
Brief Title: PrognostIc and Predictive Factors in Unresectable Locally Advanced NEC and MANEC
Acronym: NIRVANA
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1476
Record Dates: First submitted 2024-03-18; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-03

CONDITIONS: Neuroendocrine Carcinoma
Keywords: poorly differentiated neuroendocrine carcinoma; mixed adeno-neuroendocrine carcinoma; prognostic factor; predictive factor
MeSH Terms: conditions — Carcinoma, Neuroendocrine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — tumor tissue samples, peripheral blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- unresectable locally advanced neuroendocrine carcinoma: patients with extra-pulmonary, advanced neuroendocrine carcinomas
- mixed Adeno-neuroendocrine carcinomas: composed at least by 30% of a neuroendocrine (NE) and a non-neuroendocrine (non-NE) component based on the 2019 World Health Organization (WHO) classification

SUMMARY:
Extra-pulmonary (EP) poorly differentiated neuroendocrine carcinomas (NECs) represent a rare and aggressive category of neoplasms. Mixed adeno-neuroendocrine carcinomas (MANEC) are a group of rare neoplasms composed by a neuroendocrine (NE) and a non-neuroendocrine (non-NE) component, each representing at least the 30% of the neoplasm.

Considering their rarity, low prevalence and poor prognosis a clear clinical, morphological and biomolecular characterization of these neoplasms has been prevented and a clinical approach universally shared is still lacking.

DETAILED DESCRIPTION:
Extra-pulmonary (EP) poorly differentiated neuroendocrine carcinomas (NECs) represent a rare and aggressive category of neoplasms. They occur in almost 1 / 100.000 patients and the largest part is represented by gastro-entero-pancreatic (GEP) NECs (39%).

Moreover, mixed neuroendocrine non-neuroendocrine neoplasms (MiNENs) represent an even more rare entity, with a crude incidence of 0.1 / 100.000 / year, composed at least by 30% of a neuroendocrine (NE) and a non-neuroendocrine (non-NE) component based on the 2019 World Health Organization (WHO) classification. Focusing on the neuroendocrine counterpart, although the term MiNEN includes both well and poorly differentiated morphologies, the main part of them are represented by high grade neuroendocrine neoplasms categorized as MANECs in previous 2010 WHO classification that is a term still used in clinical practice is still lacking.

While for localized disease, surgery represents the cornerstone and virtually the unique curative approach, patients with metastatic disease are mostly managed with chemotherapy. Although any specific clinical practice guideline by Oncological and / or Neuroendocrine Societies has been yet developed worldwide, based on the clinical and morphological similarity with small and large cell lung NECs, cis / carbo-platinum based chemotherapy, is the most often chemotherapeutic regimen proposed in clinical practice both in NECs and MANECs from each site of origin. Other proposed options include regimens containing 5-fluorouracil/folinic-acid and irinotecan or oxaliplatin which are used also in the treatment of colo-rectal adenocarcinomas. Moreover, considering their rarity, low prevalence and poor prognosis a clear clinical, morphological and biomolecular characterization of these neoplasms has been prevented and a clinical approach universally shared is still lacking.

Therefore, a comprehensive clinical and biological characterization of these neoplasms represents an unmet medical need and a major challenge and could improve the awareness of clinicians in the management of EP-NECs and MANECs.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of unresectable locally advanced or metastatic NEC or MANEC confirmed by an expert-pathologist
* EP-primary site (included unknown primary site
* Age > 18 years
* Signed written informed consent
* Performance status ≤2
* Available tumor tissue (formalin-fixed paraffin-embedded, FFPE) (preferably within 6 months). If the tumor contained in FFPE tissue block cannot be provided in total, sections from this block should be provided that are freshly cut. Preferably, 25 slides should be provided (minimum of 15 slides). If tumor tissue is not available, patients should be willing to undergone to a new biopsy.

Exclusion Criteria:

* Diagnosis of well-differentiated NEN (G1, G2, G3)
* Collision tumors
* Cytological diagnosis of NEC or MANEC or not availability of tumor tissue for pathological analysis.
* Concurrent neoplastic disease (e.g. Advanced breast or prostatic cancer in hormonal treatment, hematologic diseases)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Extra-pulmonary (EP) poorly differentiated neuroendocrine carcinomas (NECs) and mixed neuroendocrine non-neuroendocrine neoplasms (MINENs) patients aged more than 18 years with ECOG PS minor or equal to 2.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival clinical outcome | 3 years
  The primary clinical endpoint will be the overall survival.

SECONDARY OUTCOMES:
Progression free survival clinical outcome | 3 years
  The secondary clinical endpoint will be the progression free survival
Mutational pattern | 3 years
  Mutational patterns such as BRAF, KRAS, NRAS, MSI, TP53, RB1 will be analyzed.
Prognostic and predictive factors identification | 3 years
  The progression free survival and overall survival of patients with mutations will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Spada, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No